CLINICAL TRIAL: NCT00595166
Title: Using a Sheathed Speculum to Visualize and Access the Cervix in Women With Excessive Vaginal Tissue
Status: Terminated | Type: Observational
Why Stopped: Design changed to observational, not RCT. PI left USF; study closed.
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Other Study IDs: SpecSheath
Record Dates: First submitted 2008-01-04; First posted 2008-01-16 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Healthy
Keywords: Women with excessive vaginal tissue that obstruct the examiner's view of the cervix during a vaginal speculum examination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- B: Speculum Sheath group. Participants all received the speculum sheath.
  Interventions: Device: Vaginal Speculum Sheath

INTERVENTIONS:
Device: Vaginal Speculum Sheath — Patients received the sheathed speculum exam: The clinician will begin to place the sheath onto the speculum. The sheath is attached to a thin piece of cardboard. The proximal end of the cardboard is placed between the speculum blades and is pushed toward the speculum handle. The blades of the speculum are simultaneously guided to enter the 2 pockets of the sleeve, like fingers going into a glove. The speculum exam will then be completed according to usual procedures. In the event the sheathed speculum exam is unsatisfactory the clinician will do standard of care (the clinician's usual routine at the bedside).

SUMMARY:
This new invention addresses the inadequate and incomplete visualization of the cervix in patients with excessive vaginal tissue. In general these patients are obese, or are multiparous with a history of multiple vaginal deliveries.

A vaginal speculum is a vital medical instrument that allows a health care provider to visualize the interior aspects of the vagina, as well as the distal portion of the uterus, the cervix. It is composed of 2 blades assembled together and held by a handle. The blades and the handle form a 90 degree-angle. As the user holds the handle, a lever attached to the top blade allows it to open away from the inferior blade.

When the instrument is inserted into the vagina, the two blades are separated in order to keep the anterior and posterior vaginal walls apart. In that position, the cervix and the walls of the vagina can be seen if the patient does not have an excess of loose vaginal tissue. However, in patients with excessive tissue, the sidewalls of the vagina simply collapse toward the midline between the blades because of the fact that no part of the speculum is in direct contact with the lateral walls of the vagina. This collapse prevents the complete and crucial visualization of the cervix for purposes of cervical cultures, pap smears, visual assessment of ruptured membranes, visual assessment of the degree of dilation, biopsies, and other procedures requiring access to the cervix or the uterus.

When clinicians face this dilemma, they may try the largest speculum available, and will open it as wide as possible in order to keep the lateral walls apart. Most often, they have to improvise by cutting the tip of a condom, or the thumb off a glove, or they use a sterile lateral-wall retractor. These other creative solutions can take several minutes of precious times and may still result in an inadequate visualization and suboptimal access.

A vaginal speculum sheath for retaining vaginal tissue in a lateral direction conforms to a pair of blades that are movable between an opened position and a closed position. The blades in the closed position are adapted for insertion into a vagina, and in the open position, they allow dilating the vagina in order to provide access to the cervix.

This new design includes a flexible, transparent polyurethane sleeve structure that extends between the blades when the speculum is opened. The stretched sheath is adapted to retain the lateral walls of the vagina in the open position. The elastic sleeve is designed to remain in a collapsed configuration when the blades are in a closed position to avoid interfering with insertion or withdrawal of the speculum [Reference: U.S. patent 6432048 (2002-8-13)]. Polyurethane material is FDA approved for vaginal use.

The purpose of this study is to compare standard of care speculum vs. sheathed speculum in the examination of patients with collapsing vaginal sidewalls during a gynecological speculum exam.

The primary hypothesis testing for this study will be to compare the standard of care speculum exam to a sheathed speculum exam in a prospective, randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

The following criteria must be present for randomization into the study:

Inclusion Criteria

* Age 18 to 64.
* BMI greater than 30.
* Collapsing vaginal tissue preventing the visualization of the cervix (meeting this criterion in the absence of a BMI >30 would also qualify the patient for the study).
* Able to provide written informed consent

Exclusion Criteria:

The following criteria would exclude patients from randomization into the study:

* Patients unwilling to participate in the study or provide consent.
* Presence of dyspareunia (due to chronic pelvic pain, pelvic floor dysfunction, atrophic vaginitis, or any other etiology).
* Presence of other significant pelvic pain syndromes (interstitial cystitis, endometriosis).
* Presence of active genital herpes.
* Presence of significant condyloma acuminata (may be an investigator decision).
* Any other patient deemed inappropriate for the study by the consenting or examining investigator.

Ages: 18 Years to 64 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women who were unable to have a speculum exam completed due to collapse of vaginal tissues that occludes visibility of the cervix.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2007-06; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
The main objective of the study is to assess the effectiveness of a sheathed speculum compared to standard of care procedures in providing adequate visualization and access to the cervix in patients with excessive vaginal tissue. | Once the cervix is visualized, the timing of the procedure will stop.

SECONDARY OUTCOMES:
The two speculum examination procedures will also be timed from the moment of randomization to the visualization of the cervical os. | Once the cervix is visualized, the timing of the procedure will stop.

CONTACTS AND LOCATIONS:
Overall Officials: Rony Francois, MD, PhD, Principal Investigator — University of South Florida
Locations (1):
- USF South Tampa Center for Advanced Healthcare, Tampa, Florida, United States